CLINICAL TRIAL: NCT05848830
Title: The Effects of Home-based Exercise Training and Multi-ingredient Supplementation on Functional Outcomes and Skeletal Muscle Adaptations in Patients With Myotonic Dystrophy Type 1
Brief Title: Home-based Training and Supplementation in DM1 Patients
Acronym: DM1HBET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Mark Tarnopolsky, Principal Investigator, Professor, Director of Neuromuscular and Neurometabolic Clinic, McMaster University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 15550
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Myotonic Dystrophy 1
Keywords: myotonic dystrophy, skeletal muscle, mitochondria
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Intervention Model Description: All participants will undergo 16 weeks of home-based exercise training. Half of them are randomized in an active group with a multi-ingredient supplement, and half will be given a placebo. Both the participants and the investigators are blinded to the groups.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both the participants and the investigators are blinded to the active and placebo groups. A third party, Gruppo Nutrition (Windsor, ON) will conduct the randomization for our supplemental interventions and manage blinding procedures. Neither the participants nor the investigators will be unblinded to the supplement randomization. Lastly, researchers will only be unblinded upon finishing the data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DM1 + HBEXT + MIS (Active Comparator): Participants will be asked to undergo 16 weeks of home-based training and asked to take one dose of a multi-ingredient supplement per day.
  Interventions: Dietary Supplement: Mult-ingredient supplement; Behavioral: Concurrent exercise training
- DM1 + HBEXT + PLA (Placebo Comparator): Participants will be asked to undergo 16 weeks of home-based training and asked to take one dose of a multi-ingredient supplement placebo per day.
  Interventions: Dietary Supplement: Placebo; Behavioral: Concurrent exercise training
- CONTROL (No Intervention): Healthy control subjects who will not undergo study intervention and will be used for baseline measurements and outcomes.

INTERVENTIONS:
Dietary Supplement: Mult-ingredient supplement — A mult-ingredient supplement containing Protein, both whey and casein, Creatine, Vitamin D, and Calcium. As well as antioxidants and other dietary supplements including Vitamin E, CoQ10, Alpha Lipoic Acid, L-Arginine, Beet Root Extract, Green Coffee Bean Extract, Green Tea Extract, Black Tea Extract, Curcumin, and Forskolin
  Arms: DM1 + HBEXT + MIS
Dietary Supplement: Placebo — The placebo sachet will contain micro-crystalline cellulose (inactive compound) and will be identical in look and taste to the active supplement.
  Arms: DM1 + HBEXT + PLA
Behavioral: Concurrent exercise training — All participants will undergo 16-weeks of exercise training, containing 3 days/week of resistance training and 2days/ week of aerobic training.
  Arms: DM1 + HBEXT + MIS; DM1 + HBEXT + PLA

SUMMARY:
Myotonic dystrophy type 1 (DM1) is a rare genetic disease that affects about 1 in 2100 people. Patients diagnosed with DM1 present with many symptoms, however, their muscles are mainly affected. DM1 patients experience a gradual loss of muscle, followed by an increase in body fat percentage, which makes them weaker, resulting in difficulties to perform activities of daily living, such as climbing stairs, and understandably, this affects their quality of life. DM1 currently does not have a cure. Therefore, it is very important to find ways in which we can help DM1 patients to improve their symptoms, and hopefully, improve their quality of life, and possibly improve disease prognosis. Exercise is known to improve muscle quality and function. In addition, we hypothesize that a multi-ingredient supplement (MIS) for muscle health and antioxidants for fat loss, might show improved benefits on top of exercise. Therefore, we will investigate the effects of 16-week home-based concurrent training, with MIS or placebo, on body composition, and functional measures. Lastly, we will investigate muscle adaptations in DM1 and following study intervention

DETAILED DESCRIPTION:
The present study will target patients (male and female) that have been clinically diagnosed with myotonic dystrophy type 1 with 100-1000 CTG repeats, between the ages of 19 - 60. In addition, a healthy population will serve as baseline controls, and they will be matched for age and sex, to the DM1 patients.

A total of 40 DM1 patients and 20 healthy controls will be recruited. DM1 patients will be randomized to 20 in the active group and 20 in the placebo. Both males and females will be recruited, targeting 20 males and 20 females. Corresponding 10 healthy males and 10 healthy females will be matched for sex and age, and only participate in baseline visits, measures, and sample collection.

Home-based concurrent training (HBCT) represents an exercise intervention with minimal barriers to entry. Our study will assess the effectiveness of this intervention, in combination with a multi-ingredient supplement (MIS) containing protein, creatine, antioxidants, and other dietary supplements in patients with DM1, in improving functional, clinical, and strength measures, as well as the quality of life, as assessed by scores in questionnaires. In addition, we will investigate adaptations to skeletal muscle following HBCT and MIS.

A randomized clinical trial of DM1 patients. Our study will include exercise as the over-arching intervention, with two groups nested within, DM1 patients randomized to MIS and placebo, both of which will undergo 16 weeks of home-based exercise training. Measurements and samples will be collected before and after the study intervention. A third group will include age and sex-matched healthy controls. This group will not undergo training + supplement intervention and will be used for baseline comparisons between healthy participants and DM1 patients.

Study procedures will include blood draws and muscle biopsies in each visit. In addition, participants will be asked to undergo a cardiorespiratory fitness test (VO2MAX test), a battery of functional tests (6-minute walk test, 5x sit-to-stand, one leg standing, 4-stair climb), strength testing (grip strength and knee extension tests) and lastly, clinical procedures, including ECGs and spirometry. Measurements and sample collection will be done before and after the study intervention.

ELIGIBILITY:
Age and sex-matched controls inclusion criteria:

* Healthy men and women
* Normal BMI (BMI 18.5 - 24.9 kg/m2)

Inclusion Criteria for DM1 patients:

* Male or female clinically diagnosed with DM1 (age 19 - 60 y).
* CTG repeats 100-1000.
* Normal weight (BMI 18.5 - 24.9 kg/m2) or overweight (BMI 25 - 29.9 kg/m2).
* Physically inactive (< 1 hour of formal exercise/week).
* 6-minute walk test score between 250 - 500 meters
* ECG with PR interval < 225 ms and QRS duration < 125 ms.

Exclusion Criteria for DM1 patients:

* Smoking
* Obese (BMI > 30.0 kg/m2)
* Physically active (> 1-2 hour of formal exercise/week)
* 6-minute walk test score <250 meters, chronic (> 2 weeks)
* Use of narcotic analgesic or anti-inflammatory drugs
* Type 1 or 2 diabetes (more than one anti-diabetic drug)
* Cardiovascular disease (recent myocardial infarction (< 6 months)
* Uncontrolled hypertension requiring more than 2 medications.
* Congestive heart failure requiring more than one medication for control.
* Cardiac conduction block (as above)
* Renal disease (creatinine > 140)
* Known liver disease
* Cognitive impairments limiting ability to provide informed consent
* Previous stroke with residual hemiparesis
* Active musculoskeletal injuries and/or severe osteoarthritis
* Significant weight loss in the 3-month period prior to the study
* Severe peripheral neuropathy
* Severe osteoporosis
* Use of medications known to affect protein metabolism (i.e. corticosteroids)
* Chronic obstructive or restrictive pulmonary disease (FVC < 70% of age predicted mean value)
* Asthma requiring more than two medications.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Body Composition Index | 4 months from enrolment
  Changes in ratio of fat-free mass to fat mass index as assessed via DEXA scan
VO2 Max | 4 months from enrolment
  Changes in cardiorespiratory fitness proxy measure as assessed via VO2 max testing

SECONDARY OUTCOMES:
6-minute walk test | 4 months from enrolment
  Changes in number of meters walked during the 6 minute walk test
5x sit to stand | 4 months from enrolment
  Changes in time (s) that is needed to complete 5x sit to stand from a chair
Timed up and go | 4 months from enrolment
  Changes in the time (seconds) needed to complete a timed up and go test
Leg muscle strength | 4 months from enrolment
  Changes in maximal isometric knee extension via Biodex in N*m
Grip strength | 4 months from enrolment
  Changes in grip strength (kg) using a hand dynamometer
Single leg stance test | 4 months from enrolment
  Changes in whether patients can stand on one leg for 10 s or not
Muscle fibre cross sectional area | 4 months from enrolment
  Changes in fibre cross sectional area from a muscle biopsy of vastus lateralis using immunoflourescence
Muscle stem cell mitochondrial function | 4 months from enrolment
  Changes in mitochondrial function in isolated muscle stem cells of DM1 patients via seahorse assay

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No